CLINICAL TRIAL: NCT04636112
Title: Effects of Sleep Habits on Acute Myocardial Infarction Risk and Severity of Coronary Artery Disease in Chinese Population
Brief Title: Sleep Habits and AMI and Gensini Score
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Jiangning Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Liansheng Wang, Professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: NSFC
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Sleep Disorder; Acute Myocardial Infarction
Keywords: sleep habits; sleep duration; daytime napping; Gensini score; late sleeping
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Patients hospitalized and diagnosed as non-AMI during the same time period were matched. All patients underwent coronary angiography and CAD was defined as at least one main coronary artery with > 50% narrowing of luminal diameter.
- AMI group: Patients were diagnosed as MI when a cardiac biomarker (preferably cardiac troponin) rose or fell at least one value in its 99th percentile upper reference limit and at least one of the following criteria was met, including ischemic symptoms, electrocardiogram (ECG) changes of new ischemia, pathologic Q waves in the ECG, imaging evidence of new loss of viable myocardium or new regional wall motion abnormality, identification of an intracoronary thrombus by angiography or autopsy.

SUMMARY:
This study was to examine the effects of sleep habits on acute myocardial infarction (AMI) risk and severity of coronary artery disease (CAD) in Chinese population from two centers. A total of 873 patients were recruited from the inpatient cardiology department of the Affiliated Jiangning Hospital and the First Affiliated Hospital of Nanjing Medical University. Investigators used a 17-item sleep factors questionnaire (SFQ) to evaluate sleep habits comprehensively by face-to-face interview.

DETAILED DESCRIPTION:
Growing evidence indicates that poor sleep harms health. Early to bed and early to rise is considered as a healthy lifestyle in Chinese population. The current study aimed to examine the effects of sleep habits on acute myocardial infarction (AMI) risk and severity of coronary artery disease (CAD) in Chinese population from two centers. A total of 873 patients including 314 with AMI were recruited from the inpatient cardiology department of the Affiliated Jiangning Hospital and the First Affiliated Hospital of Nanjing Medical University. 559 controls included 395 CAD cases and 164 non-CAD cases. Investigators used a 17-item sleep factors questionnaire (SFQ) to evaluate sleep habits comprehensively by face-to-face interview. The severity of CAD was assessed by Gensini score in AMI and CAD groups. The effects of sleep factors on AMI risk and Gensini score were examined by unconditional logistic regression. The timing of sleep (24:00 and after), sleep duration (<6h) and frequency of night-time waking (3 times) increased the risk of AMI. In subjects with age ≤60 years, daytime napping reduced the risk of AMI. The correlation between sleep quality and AMI became insignificant after subgroup analysis by age. Short sleep duration also increased the risk of high Gensini score.

ELIGIBILITY:
Inclusion Criteria:

1. underwent coronary angiography;
2. can complete sleep factors questionnaire.

Exclusion Criteria:

1. mental diseases;
2. sleep apnea;
3. chronic obstructive pulmonary disease;
4. stroke sequelae;
5. arthritis;
6. renal failure;
7. tumor and a history of revascularization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A case-control study was designed to investigate the effects of sleep habits on AMI and severity of CAD. After patients were in stable condition, trained physicians administered a questionnaire survey by a face-to-face interview. Information on demographic characteristics, hypertension, diabetes and dyslipidemia history, drug use, smoking, drinking, dietary habits, exercise and sleep habits were collected.
Sampling Method: Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
a 17-item sleep factors questionnaire | in the last year before enrollment
  SFQ included sleep quality, sleep duration at night, timing of sleep and waking up, insomnia and night-time waking frequency, sleep medication use, night work, daytime napping, light at night (LAN) exposure and sleep noise.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Liansheng, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson NF, Badr MS, Belenky G, Bliwise DL, Buxton OM, Buysse D, Dinges DF, Gangwisch J, Grandner MA, Kushida C, Malhotra RK, Martin JL, Patel SR, Quan SF, Tasali E. Recommended Amount of Sleep for a Healthy Adult: A Joint Consensus Statement of the American Academy of Sleep Medicine and Sleep Research Society. Sleep. 2015 Jun 1;38(6):843-4. doi: 10.5665/sleep.4716. PMID 26039963
- [Background] Buxton OM, Marcelli E. Short and long sleep are positively associated with obesity, diabetes, hypertension, and cardiovascular disease among adults in the United States. Soc Sci Med. 2010 Sep;71(5):1027-36. doi: 10.1016/j.socscimed.2010.05.041. Epub 2010 Jun 16. PMID 20621406
- [Background] Nuyujukian DS, Beals J, Huang H, Johnson A, Bullock A, Manson SM, Jiang L; Special Diabetes Program for Indians Diabetes Prevention Demonstration Project. Sleep Duration and Diabetes Risk in American Indian and Alaska Native Participants of a Lifestyle Intervention Project. Sleep. 2016 Nov 1;39(11):1919-1926. doi: 10.5665/sleep.6216. PMID 27450685
- [Background] Kobayashi D, Takahashi O, Deshpande GA, Shimbo T, Fukui T. Association between weight gain, obesity, and sleep duration: a large-scale 3-year cohort study. Sleep Breath. 2012 Sep;16(3):829-33. doi: 10.1007/s11325-011-0583-0. Epub 2011 Sep 3. PMID 21892668
- [Background] Kim JY, Yadav D, Ahn SV, Koh SB, Park JT, Yoon J, Yoo BS, Lee SH. A prospective study of total sleep duration and incident metabolic syndrome: the ARIRANG study. Sleep Med. 2015 Dec;16(12):1511-5. doi: 10.1016/j.sleep.2015.06.024. Epub 2015 Sep 28. PMID 26611949
- [Background] Thomson CA, Morrow KL, Flatt SW, Wertheim BC, Perfect MM, Ravia JJ, Sherwood NE, Karanja N, Rock CL. Relationship between sleep quality and quantity and weight loss in women participating in a weight-loss intervention trial. Obesity (Silver Spring). 2012 Jul;20(7):1419-25. doi: 10.1038/oby.2012.62. Epub 2012 Mar 8. PMID 22402738
- [Background] Cappuccio FP, Stranges S, Kandala NB, Miller MA, Taggart FM, Kumari M, Ferrie JE, Shipley MJ, Brunner EJ, Marmot MG. Gender-specific associations of short sleep duration with prevalent and incident hypertension: the Whitehall II Study. Hypertension. 2007 Oct;50(4):693-700. doi: 10.1161/HYPERTENSIONAHA.107.095471. Epub 2007 Sep 4. PMID 17785629
- [Background] Cappuccio FP, Cooper D, D'Elia L, Strazzullo P, Miller MA. Sleep duration predicts cardiovascular outcomes: a systematic review and meta-analysis of prospective studies. Eur Heart J. 2011 Jun;32(12):1484-92. doi: 10.1093/eurheartj/ehr007. Epub 2011 Feb 7. PMID 21300732
- [Background] Campos H, Siles X. Siesta and the risk of coronary heart disease: results from a population-based, case-control study in Costa Rica. Int J Epidemiol. 2000 Jun;29(3):429-37. PMID 10869314
- [Background] Sharma M, Sawhney JP, Panda S. Sleep quality and duration - potentially modifiable risk factors for Coronary Artery Disease? Indian Heart J. 2014 Nov-Dec;66(6):565-8. doi: 10.1016/j.ihj.2014.10.412. Epub 2014 Nov 4. PMID 25634385
- [Background] Xie D, Li W, Wang Y, Gu H, Teo K, Liu L, Yusuf S; INTERHEART China study Investigators. Sleep duration, snoring habits and risk of acute myocardial infarction in China population: results of the INTERHEART study. BMC Public Health. 2014 May 29;14:531. doi: 10.1186/1471-2458-14-531. PMID 24885282
- [Background] Wang D, Ruan W, Chen Z, Peng Y, Li W. Shift work and risk of cardiovascular disease morbidity and mortality: A dose-response meta-analysis of cohort studies. Eur J Prev Cardiol. 2018 Aug;25(12):1293-1302. doi: 10.1177/2047487318783892. Epub 2018 Jun 22. PMID 29929393
- [Background] Sinning C, Lillpopp L, Appelbaum S, Ojeda F, Zeller T, Schnabel R, Lubos E, Jagodzinski A, Keller T, Munzel T, Bickel C, Blankenberg S. Angiographic score assessment improves cardiovascular risk prediction: the clinical value of SYNTAX and Gensini application. Clin Res Cardiol. 2013 Jul;102(7):495-503. doi: 10.1007/s00392-013-0555-4. Epub 2013 Mar 23. PMID 23519584
- [Background] Yang WS, Fu WX, Wang X, Deng Q, Wang L, Wang LY, Zhao H, Fan WY, Huang SX. Comprehensive assessments of long-term sleep habits in epidemiological study: Validity and reliability of sleep factors questionnaire (SFQ) among Chinese women. J Psychosom Res. 2017 Apr;95:12-18. doi: 10.1016/j.jpsychores.2017.02.005. Epub 2017 Feb 10. PMID 28314544
- [Background] Taheri S, Lin L, Austin D, Young T, Mignot E. Short sleep duration is associated with reduced leptin, elevated ghrelin, and increased body mass index. PLoS Med. 2004 Dec;1(3):e62. doi: 10.1371/journal.pmed.0010062. Epub 2004 Dec 7. PMID 15602591
- [Background] Stang A, Dragano N, Moebus S, Mohlenkamp S, Schmermund A, Kalsch H, Erbel R, Jockel KH; Heinz Nixdorf Recall Investigative Group. Midday naps and the risk of coronary artery disease: results of the Heinz Nixdorf Recall Study. Sleep. 2012 Dec 1;35(12):1705-12. doi: 10.5665/sleep.2248. PMID 23204613
- [Background] Merikanto I, Lahti T, Puolijoki H, Vanhala M, Peltonen M, Laatikainen T, Vartiainen E, Salomaa V, Kronholm E, Partonen T. Associations of chronotype and sleep with cardiovascular diseases and type 2 diabetes. Chronobiol Int. 2013 May;30(4):470-7. doi: 10.3109/07420528.2012.741171. Epub 2013 Jan 2. PMID 23281716